CLINICAL TRIAL: NCT04417751
Title: Care at 360º: A Long-term Individual Cognitive Stimulation Program for Older Adults With Neurocognitive Disorders, Non-Institutionalized and Socially Vulnerable
Brief Title: Care at 360º: A Long-term Individual Cognitive Stimulation Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CEDIARA - Assoc. Solidariedade Social de Ribeira de Fráguas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 23052020
Record Dates: First submitted 2020-05-27; First posted 2020-06-05 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2020-07

CONDITIONS: Neurocognitive Disorders; Dementia; Cognitive Impairment; Cognitive Decline; Cognitive Dysfunction; Social Behavior
Keywords: older adults; cognitive stimulation; dementia; intervention; cognition; individual intervention; social vulnerability; quality of life; aged; non-pharmacological therapy; neurocognitive disorder; psychosocial
MeSH Terms: conditions — Neurocognitive Disorders; Dementia; Cognitive Dysfunction; Social Behavior

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Intervention group will receive 47 sessions of individual CS and participate in 3 evaluation sessions. The CS program will last 1 year and each individual CS session will last approximately 45 minutes.
  Interventions: Behavioral: Cognitive Stimulation
- Control Group (No Intervention): Participants assigned to the control group will maintain their usual treatment in the institution, participating in the activities previously assigned to their individual care plan.

INTERVENTIONS:
Behavioral: Cognitive Stimulation — The intervention includes 50 sessions, over the course of one year, being that 3 of those sessions will be the pretest, intratest and posttest evaluations. The intervention sessions will last approximately 45 minutes and they will be developed according to the following structure: welcoming and greeting the participants (5 minutes); reality orientation therapy (10 minutes), cognitive stimulation [CS] activity (25 minutes); return to calm and closure of the session, and session evaluation (5 minutes). CS sessions will be conducted in an individual intervention format. The intervention sessions will include several activities based on different non-pharmacological therapies (e.g., reminiscence therapy, reality orientation therapy, cognitive training) whose effectiveness in older adults with neurocognitive disorders has been scientifically proven. All individual CS sessions will be conducted by one therapist (clinical psychologist) with more than five years of experience in CS.
  Arms: Intervention Group

SUMMARY:
The aim of the intervention proposed in the present study is to assess the effect of a cognitive stimulation (CS) intervention program in an individual and long-term format, for non-institutionalized elderly people with neurocognitive disorders and in a situation of social vulnerability. Specifically, to test the effectiveness of CS on the global cognitive state, on mood state, on quality of life and on functional state. The program will be composed by 50 sessions, including three of assessment sessions (pre, intra and post-intervention). Each session will have a duration of 45 minutes with a weekly frequency. Control group participants will maintain their treatment as usual.

DETAILED DESCRIPTION:
According to World Health Organization, between 2000 and 2050, the proportion of the planet's inhabitants over 60 years of age will double, from 11% to 22%. Specifically, this age group will increase from 605 million to 2000 million worldwide by the middle of the century.

As for Portugal, according to data from the National Statistics Institute, the resident population was composed by 21.5% of elderly people. This percentage was higher than the European Union average of 28 countries (EU28), which does not reach 20%, with Portugal being the fourth country with the highest percentage of elderly people.

Aging implies an increased risk for the development of biological, socioeconomic and psychosocial vulnerabilities, derived from biological decline and from an increase in pathologies associated with aging itself. In view of the current Covid-19 pandemic, the risk of vulnerability is heightened.

There are several chronic diseases that affect the elderly. Regarding mental disorders, the most frequent as age, are neurocognitive disorders. The diagnostic criteria for this pathology emphasize cognitive changes, and as such, it is clinically based on cognitive and memory decline.

There is evidence that in the early stages of neurocognitive disorders, people are able to learn and improve their cognitive function through interventions, such as cognitive stimulation. There are three types of cognitive intervention: cognitive stimulation, cognitive rehabilitation and cognitive training. Cognitive rehabilitation is an individual approach to cognitive impairment and improves daily functioning. Cognitive training is designed for the patient to perform a set of tasks in order to improve or maintain cognitive function through guided practice. Cognitive stimulation is an intervention where the cognitive domains are not used isolated, but rather integrated. Cognitive stimulation can be structured in an individual or group format. Individual cognitive stimulation includes activities designed to stimulate cognition, conducted only with the therapist and the patient.

In a Portuguese study, with participants in the same geographic area, who applied individual cognitive stimulation therapy to patients with mild neurocognitive disorder, over a year, a significant improvement was found in the intervention group in terms of cognitive performance and a reduction of depressive symptoms, with a moderate to large effect size, suggesting that cognitive stimulation therapy is effective in an individual format.

According to this evidence, the National Institute for Health and Clinical Excellence recommended cognitive stimulation as a non-pharmacological therapy for people with mild to moderate neurocognitive disorder.

In a systematic review about cognitive stimulation, studies showed a strong evidence that cognitive stimulation has a positive impact on cognitive performance, depression, activities of daily living and behavior in people with neurocognitive disorders.

Considering the previous information, the aim of this project is to apply cognitive stimulation in an individual format to improve cognitive status and performance, quality of life and functionality, and reduce depressive symptoms in non-institutionalized elderly people in a vulnerable social context with a diagnosis of neurocognitive disorder.

ELIGIBILITY:
Inclusion Criteria:

* Being flagged as a person in a socially vulnerable context.
* Being 65 years of age or over.
* Having a neurocognitive disorder according to the diagnostic criteria of the Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-5) (2014).
* Being a native Portuguese speaker.
* Residing in the region of Ribeira de Fráguas.

Exclusion Criteria:

* Not having preserved the ability to communicate and understand.
* To suffer from a severe or acute illness that makes the participation in the sessions impossible.
* Presence of severe neuropsychiatric symptoms that prevent participation in the sessions or uncontrolled psychotic conditions.
* Being institutionalized.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 59 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-07-26 (Actual); Study Completion 2021-07-26 (Actual)

PRIMARY OUTCOMES:
Cognitive state evaluated through Mini-Mental State Examination | Pre-intervention
  Significant statistic improvement in the participant's test scores between pre-intervention, intra-intervention and postintervention assessments. Mini-Mental State Examination is a brief screening test for cognitive function. Assesses 6 cognitive functions: orientation, registration, attention and calculation, recall, language and visuoconstructive ability.
  Global score ranges from 0-30 points, higher scores indicate better cognitive function.
Change in cognitive state evaluated through Mini-Mental State Examination | 6 months after the beginning of the intervention
  Significant statistic improvement in the participant's test scores between pre-intervention, intra-intervention and postintervention assessments. Mini-Mental State Examination is a brief screening test for cognitive function. Assesses 6 cognitive functions: orientation, registration, attention and calculation, recall, language and visuoconstructive ability.
  Global score ranges from 0-30 points, higher scores indicate better cognitive function.
Change in cognitive state evaluated through Mini-Mental State Examination | 12 months after the beginning of the intervention
  Significant statistic improvement in the participant's test scores between pre-intervention, intra-intervention and postintervention assessments. Mini-Mental State Examination is a brief screening test for cognitive function. Assesses 6 cognitive functions: orientation, registration, attention and calculation, recall, language and visuoconstructive ability.
  Global score ranges from 0-30 points, higher scores indicate better cognitive function.
Cognitive performance evaluated through Montreal Cognitive Assessment | Pre-intervention
  It's a 32-item mild cognitive impairment screening instrument that assesses eight cognitive functions: visuospatial/executive, naming, memory, attention, language, abstraction, delayed recall and orientation. Montreal Cognitive Assessment score is calculated by adding the points of the tasks successfully completed, and it ranges from 0 to 30 points, being that higher scores indicate better cognitive performance.
Change in cognitive performance evaluated through Montreal Cognitive Assessment | 6 months after the beginning of the intervention
  It's a 32-item mild cognitive impairment screening instrument that assesses eight cognitive functions: visuospatial/executive, naming, memory, attention, language, abstraction, delayed recall and orientation. Montreal Cognitive Assessment score is calculated by adding the points of the tasks successfully completed, and it ranges from 0 to 30 points, being that higher scores indicate better cognitive performance.
Change in cognitive performance evaluated through Montreal Cognitive Assessment | 12 months after the beginning of the intervention
  It's a 32-item mild cognitive impairment screening instrument that assesses eight cognitive functions: visuospatial/executive, naming, memory, attention, language, abstraction, delayed recall and orientation. Montreal Cognitive Assessment score is calculated by adding the points of the tasks successfully completed, and it ranges from 0 to 30 points, being that higher scores indicate better cognitive performance.

SECONDARY OUTCOMES:
Depressive symptoms evaluated through Geriatric Depression Scale -15 | Pre intervention
  Significant statistic improvement in the participant's test scores between pre-intervention, intra-intervention and postintervention assessments. Geriatric Depression Scale -15 is a screening test for depressive symptoms in elderly adults. Assesses depression in the elderly by distinguishing between depressive and dementia symptoms. This instrument does not include somatic conditions common to the elderly, such as appetite, sleep or sexual disturbances, or lower energy level. The overall score ranges from 0 to 15. The higher the score, the greater the severity of the depressive symptoms.
Change in depressive symptoms evaluated through Geriatric Depression Scale -15 | 6 months after the beginning of the intervention
  Significant statistic improvement in the participant's test scores between pre-intervention, intra-intervention and postintervention assessments. Geriatric Depression Scale -15 is a screening test for depressive symptoms in elderly adults. Assesses depression in the elderly by distinguishing between depressive and dementia symptoms. This instrument does not include somatic conditions common to the elderly, such as appetite, sleep or sexual disturbances, or lower energy level. The overall score ranges from 0 to 15. The higher the score, the greater the severity of the depressive symptoms.
Change in depressive symptoms evaluated through Geriatric Depression Scale -15 | 12 months after the beginning of the intervention
  Significant statistic improvement in the participant's test scores between pre-intervention, intra-intervention and postintervention assessments. Geriatric Depression Scale -15 is a screening test for depressive symptoms in elderly adults. Assesses depression in the elderly by distinguishing between depressive and dementia symptoms. This instrument does not include somatic conditions common to the elderly, such as appetite, sleep or sexual disturbances, or lower energy level. The overall score ranges from 0 to 15. The higher the score, the greater the severity of the depressive symptoms.
Quality of life evaluated through Quality of Life - Alzheimer's Disease: score | Pre-intervention
  Significant statistic improvement in the participant's test scores between pre-intervention assessment and postintervention assessment. Quality of Life - Alzheimer's Disease is an instrument to assess quality of life in people diagnosed with dementia, gathering information from the patient and the caregiver. It is composed by 13 items regarding perception of health, mood, functional abilities, interpersonal relationships and hobbies, decision making ability and life in general. It has good psychometric characteristics and it's use has been recommended to evaluate psychosocial interventions. Scores range between 13 - 52 points. Higher scores indicate better quality of life.
Change in quality of life evaluated through Quality of Life - Alzheimer's Disease: score | 6 months after the beginning of the intervention
  Significant statistic improvement in the participant's test scores between pre-intervention assessment and postintervention assessment. Quality of Life - Alzheimer's Disease is an instrument to assess quality of life in people diagnosed with dementia, gathering information from the patient and the caregiver. It is composed by 13 items regarding perception of health, mood, functional abilities, interpersonal relationships and hobbies, decision making ability and life in general. It has good psychometric characteristics and it's use has been recommended to evaluate psychosocial interventions. Scores range between 13 - 52 points. Higher scores indicate better quality of life.
Change in quality of life evaluated through Quality of Life - Alzheimer's Disease: score | 12 months after the beginning of the intervention
  Significant statistic improvement in the participant's test scores between pre-intervention assessment and postintervention assessment. Quality of Life - Alzheimer's Disease is an instrument to assess quality of life in people diagnosed with dementia, gathering information from the patient and the caregiver. It is composed by 13 items regarding perception of health, mood, functional abilities, interpersonal relationships and hobbies, decision making ability and life in general. It has good psychometric characteristics and it's use has been recommended to evaluate psychosocial interventions. Scores range between 13 - 52 points. Higher scores indicate better quality of life.
Functional status is assessed using the Lawton and Brody Instrumental Activities of Daily Living. | Pre-intervention
  It's an instrument that assesses the independence level of the elderly people regarding IADL's. A score is assigned according to the person's ability to perform a given task. A set of three, four or five options is suggested for each question, which is scored from 1 to 3, 1 to 4 or 1 to 5 points. The highest score corresponds to a greater degree of dependency. If a task does not apply because the person did not perform it in the pre-morbid period, the score for that task is not included in the total score, that is, the maximum possible score includes only the maximum scores of the tasks that the person performed. The score ranges from 8 to 30 points (a score of 8 points means that th person is independent; between 9 and 20 points means a moderate dependency; greater than 20 points means severe dependency).
Change in functional status is assessed using the Lawton and Brody Instrumental Activities of Daily Living. | 6 months after the beginning of the intervention
  It's an instrument that assesses the independence level of the elderly people regarding IADL's. A score is assigned according to the person's ability to perform a given task. A set of three, four or five options is suggested for each question, which is scored from 1 to 3, 1 to 4 or 1 to 5 points. The highest score corresponds to a greater degree of dependency. If a task does not apply because the person did not perform it in the pre-morbid period, the score for that task is not included in the total score, that is, the maximum possible score includes only the maximum scores of the tasks that the person performed. The score ranges from 8 to 30 points (a score of 8 points means that th person is independent; between 9 and 20 points means a moderate dependency; greater than 20 points means severe dependency).
Change in functional status is assessed using the Lawton and Brody Instrumental Activities of Daily Living. | 12 months after the beginning of the intervention
  It's an instrument that assesses the independence level of the elderly people regarding IADL's. A score is assigned according to the person's ability to perform a given task. A set of three, four or five options is suggested for each question, which is scored from 1 to 3, 1 to 4 or 1 to 5 points. The highest score corresponds to a greater degree of dependency. If a task does not apply because the person did not perform it in the pre-morbid period, the score for that task is not included in the total score, that is, the maximum possible score includes only the maximum scores of the tasks that the person performed. The score ranges from 8 to 30 points (a score of 8 points means that th person is independent; between 9 and 20 points means a moderate dependency; greater than 20 points means severe dependency).

OTHER OUTCOMES:
Sociodemographic data collected through a sociodemographic questionnaire | Pre-intervention
  Sociodemographic data will be collected using a sociodemographic questionnaire, designed specifically for this study, regarding information about age, gender, literacy, health conditions, among others.
Adherence to the intervention and dropouts evaluated through a session form | [Pre, intra (6 months) and post intervention (12 months)]
  Adherence to the intervention and dropouts will be assessed using a session form, designed specifically for this study, completed by the technician after each session, regarding the attendance and mood/behavior of the participants throughout the intervention sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Susana I Justo Henriques, PhD, Principal Investigator — Health Sciences Research Unit: Nursing (UICISA: E), ESEnfC; Ana E Marques Castro, MSc, Principal Investigator — CEDIARA - Assoc. Solidariedade Social de Ribeira de Fráguas; Enrique Pérez Sáez, PhD, Principal Investigator — National Reference Centre for Alzheimer's and Dementia Care, Imserso
Locations (1):
- Cediara - Social Solidarity Association of Ribeira de Fráguas, Ribeira de Fráguas, Albergaria-a-Velha, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Apóstolo JLA, Bobrowicz-Campos EM, Reis, IAC, Henriques SJ., Correia CAV. Exploring the screening capacity of the European Portuguese version of the 15-item Geriatric Depression Scale. Revista de Psicopatología y Psicología Clínica. 2018; 23(2): 99-107. https://doi.org/10.5944/rppc.vol.23.num.2.2018.21050
- [Background] Apóstolo JL, Loureiro LMJ, Carvalho IA, Alves I, Batista DF, Sfetcu R. Contribution to the adaptation of the Geriatric Depression Scale-15 into Portuguese. Revista de Enfermagem Referencia. 2014; IV(3): 65-73. https://doi.org/10.12707/RIV14033
- [Background] Barrios H, Verdelho A, Narciso S, Goncalves-Pereira M, Logsdon R, de Mendonca A. Quality of life in patients with cognitive impairment: validation of the Quality of Life-Alzheimer's Disease scale in Portugal. Int Psychogeriatr. 2013 Jul;25(7):1085-96. doi: 10.1017/S1041610213000379. Epub 2013 Mar 27. PMID 23534370
- [Background] Clare L, Woods RT. Cognitive training and cognitive rehabilitation for people with early-stage Alzheimer's disease: A review. Neuropsychological Rehabilitation. 2004; 14: 385-401. https://doi.org/10.1080/09602010443000074
- [Background] Clare L, Wilson BA, Carter G, Breen K, Gosses A, Hodges JR. Intervening with everyday memory problems in dementia of Alzheimer type: an errorless learning approach. J Clin Exp Neuropsychol. 2000 Feb;22(1):132-46. doi: 10.1076/1380-3395(200002)22:1;1-8;FT132. PMID 10649552
- [Background] Davis RN, Massman PJ, Doody RS. Cognitive intervention in Alzheimer disease: a randomized placebo-controlled study. Alzheimer Dis Assoc Disord. 2001 Jan-Mar;15(1):1-9. doi: 10.1097/00002093-200101000-00001. PMID 11236819
- [Background] Filipin F, Feldman M, Taragano FE, Martelli M, Sánchez V, García V, … Dillon C. The efficacy of cognitive stimulation on depression and cognition in elderly patients with cognitive impairment: A retrospective cohort study. AIMS Medical Science. 2015; 3(1): 1-14. https://doi.org/10.3934/medsci.2016.1.1
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Freitas S, Simoes MR, Alves L, Santana I. The Relevance of Sociodemographic and Health Variables on MMSE Normative Data. Appl Neuropsychol Adult. 2015;22(4):311-9. doi: 10.1080/23279095.2014.926455. Epub 2014 Dec 22. PMID 25531579
- [Background] Guerreiro M, Silva AP, Botelho MA, Leitão O, Castro-Caldas A, Garcia C. Adaptação à população portuguesa da tradução do Mini Mental State Examination (MMSE). Revista Portuguesa de Neurologia. 1994; 1: 9-10.
- [Background] Justo-Henriques SI, Marques-Castro AE, Otero P, Vazquez FL, Torres AJ. [Long-term individual cognitive stimulation program in patients with mild neurocognitive disorder: a pilot study]. Rev Neurol. 2019 Apr 1;68(7):281-289. doi: 10.33588/rn.6807.2018321. Spanish. PMID 30906977
- [Background] Lawton MP, Brody EM. Assessment of older people: self-maintaining and instrumental activities of daily living. Gerontologist. 1969 Autumn;9(3):179-86. No abstract available. PMID 5349366
- [Background] Lobbia A, Carbone E, Faggian S, Gardini S, Piras F, Spector E, Borella E. The efficacy of cognitive stimulation therapy (CST) for people with mild-to-moderate dementia: A review. European Psychologist. 2018; 24(3): 257-277. https://doi.org/10.1027/1016-9040/a000342
- [Background] Loewenstein DA, Acevedo A, Czaja SJ, Duara R. Cognitive rehabilitation of mildly impaired Alzheimer disease patients on cholinesterase inhibitors. Am J Geriatr Psychiatry. 2004 Jul-Aug;12(4):395-402. doi: 10.1176/appi.ajgp.12.4.395. PMID 15249277
- [Background] Logsdon RG, Gibbons LE, McCurry SM, Teri L. Quality of life in Alzheimer's disease: Patient and caregiver reports. Journal of Mental Health and Aging. 1999; 5: 21-32.
- [Background] Moniz-Cook E, Vernooij-Dassen M, Woods R, Verhey F, Chattat R, De Vugt M, Mountain G, O'Connell M, Harrison J, Vasse E, Droes RM, Orrell M; INTERDEM group. A European consensus on outcome measures for psychosocial intervention research in dementia care. Aging Ment Health. 2008 Jan;12(1):14-29. doi: 10.1080/13607860801919850. PMID 18297476
- [Background] Morgado J, Rocha CS, Maruta C, Guerreiro M, Martins IP. Novos valores normativos do Mini-Mental Sate Examination. Sinapse. 2009; 2: 10-16.
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Rodrigues NO, Neri AL. [Social, individual and programmatic vulnerability among the elderly in the community: data from the FIBRA Study conducted in Campinas, Sao Paulo, Brazil]. Cien Saude Colet. 2012 Aug;17(8):2129-39. doi: 10.1590/s1413-81232012000800023. Portuguese. PMID 22899153
- [Background] Sheikh JI, Yesavage JA. Geriatric depression scale (GDS): Recent evidence and development of a shorter version. Clinical Gerontologist. 1986; 5(1-2): 165-173. https://doi.org/10.1300/j018v05n01_09
- [Background] Wilson B. Towards a comprehensive model of cognitive rehabilitation. Neuropsychological Rehabilitation. 2002; 12(2): 97-110. https://doi.org/10.1080/09602010244000020
- [Background] Woods B, Aguirre E, Spector AE, Orrell M. Cognitive stimulation to improve cognitive functioning in people with dementia. Cochrane Database Syst Rev. 2012 Feb 15;(2):CD005562. doi: 10.1002/14651858.CD005562.pub2. PMID 22336813
- [Derived] Justo-Henriques SI, Perez-Saez E, Marques-Castro AE, Carvalho JO. Effectiveness of a year-long individual cognitive stimulation program in Portuguese older adults with cognitive impairment. Neuropsychol Dev Cogn B Aging Neuropsychol Cogn. 2023 May;30(3):321-335. doi: 10.1080/13825585.2021.2023458. Epub 2022 Jan 11. PMID 35012439